CLINICAL TRIAL: NCT06885398
Title: Intra-Arrest-Ventilation - a Prospective Randomized Trial in Human Cadavers II
Brief Title: Intra Arrest Ventilation in Human Cadavers II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muehlenkreiskliniken, MKK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1341
Record Dates: First submitted 2025-02-26; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Ventilation During Resuscitation
Keywords: Cardiac arrest; Airway management; Cadaver; Heart diseases; Heart arrest; Death; cardiovascular diseases
MeSH Terms: conditions — Heart Arrest; Cadaver; Heart Diseases; Death; Cardiovascular Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BIPAP (Bi-Level positive airway pressure) (Active Comparator)
  Interventions: Other: treatment
- CPAP ASB (continouos positive airway pressure with assisted spontaneous breathing) (Active Comparator)
  Interventions: Other: treatment
- CCSV (Chest Compression Synchronized Ventilation) (Active Comparator)
  Interventions: Other: treatment

INTERVENTIONS:
Other: treatment — * Endotracheal Tube Ventilation with an endotracheal tub
  * Laryngeal tube Ventilation with a laryngeal tube
  * Laryngeal mask Ventilation with a laryngeal mask
  * I-Gel-Laryngeal Mask Ventilation with an I-Gel-laryngeal mask

SUMMARY:
The study investigates the influence of three types of ventilation mode by using Bi-Level positive airway pressure (pinsp 20 mbar, PEEP 5, AF 10/min) with two different types of ventilators ( Medumat vs. MeduVENT ), Continuous positive airway pressure (PEEP 5, AF 10/min, ASB 10) and Chest Compression Synchronized Ventilation (pInsp = 30 vs. 60 mbar; respiratory rate = chest compression rate, PEEP 5) with regard to achieving a sufficient tidal volume and the tightness of various supraglottic airway devices (laryngeal mask, i-Gel-laryngeal mask, laryngeal tube) and endotracheal intubation.

DETAILED DESCRIPTION:
The European Resuscitation Council (ERC) guidelines for cardiopulmonary resuscitation (CPR) recommend uninterrupted chest compressions and continuous ventilation as soon as a patient is endotracheally intubated or a supraglottic airway (SGA) is positioned.

Recently, SGAs have been adopted by emergency medical services worldwide as the primary tool for airway management during CPR. SGAs offer limited protection against aspiration compared to endotracheal intubation (ETI) and may increase the risk of aspiration. A new ventilation mode (Chest Compression Synchronized Ventilation [CCSV]) is now available for resuscitation with uninterrupted chest compressions.

The study investigates the influence of three types of ventilation mode by using Bi-Level positive airway pressure with two kind ventilators (pinsp 20 mbar, PEEP 5, AF 10/min), Continuous positive airway pressure (PEEP 5, AF 10/min, ASB 10) and Chest Compression Synchronized Ventilation (pInsp = 30 vs. 60 mbar; respiratory rate = chest compression rate, PEEP 5) with regard to achieving a sufficient tidal volume and the tightness of various supraglottic airway devices (laryngeal mask, i-Gel-laryngeal mask, laryngeal tube) and endotracheal intubation.

Gender, age, height and weight are documented (external post-mortem examination). The respective body donor is randomly assigned to a group. The grouping determines the order in which the means of airway management (SGA, ETI) are used.

Initial airway management is performed with an ETI with blockage of 40 mmH2O). The body donor is then bronchoscoped. A gastric tube is placed and the pressure probe to be used is calibrated if necessary. Positive pressure ventilation (pInsp = 35 mbar, positive end-expiratory pressure (PEEP) = 12 mbar, frequency = 10 min-1) is performed for 2 minutes to recruit the lungs. Vt is documented.

Mechanical cardiopulmonary resuscitation (CPR) is then performed for minutes (4 cycles) using the mechanical chest compression device in accordance with ERC 2015. Ventilation pressure and flow curves are continuously recorded by the respirator (Medumat Standard² and MeduVENT by the company Weinmann GmbH). Leaks are detected via the automatically initiated ventilation curves, measured and recorded by the ventilator. Ventilation takes place for 4 minutes with CPAP ASB, 4 minutes in BIPAP mode with Medumat, 4 minutes with MeduVENT and 4 minutes in CCSV mode with an pinsp of 30 and 4 minutes with 60 mbar . At the end of the cycle, the body donor is intubated with one of the remaining airway devices, and the lungs are recruited again and mechanical CPR is performed again for 20 minutes using the 3 ventilation modes. All in all the time durance of CPR for one donor will be 100 minutes by using all four airway devices.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years of age

Exclusion Criteria:

* Adult respiratory distress syndrome (ARDS)
* Severe lung or thoracic injuries
* Pneumothorax
* Abnormal airways
* Tracheostoma
* severe aspirations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
gained tidalvolume with different airway devices in BIPAP | After beginning of ventilation up to 4 minutes each device
  mean expiratory volume compared to ideal tidalvolume gained by using different airway devices in BIPAP
gained ventilation volume with different airway devices in CPAP-ASB | After beginning of ventilation up to 4 minutes each device
  mean ventilation volume compared to ideal ventilation volume gained by using different airway devices in CPAP-ASB
occurred ventilation pressure with different airway devices in CCSV | After beginning of ventilation up to 4 minutes each device
  mean ventilation pressure needed to develope a sufficient tidalvolume by using different airway devices in CCSV

SECONDARY OUTCOMES:
Mean peak pressure | After beginning of ventilation up to 4 minutes each device
  Mean peak pressure during ventilation
Inspiratory pressure | After beginning of ventilation up to 4 minutes each device
  Inspiratory pressure during ventilation
Peak pressure | After beginning of ventilation up to 4 minutes each device
  Peak pressure during ventilation
Leakage volume | After beginning of ventilation up to 4 minutes each device
  Leakage volume during ventilation
Respiratory Rate | After beginning of ventilation up to 4 minutes each device
  Respiratory Rate during ventilation

IPD SHARING:
Plan to Share IPD: No